CLINICAL TRIAL: NCT06643130
Title: A Multi-center, Randomized, Double-blind, Parallel, Phase Ⅲ Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of JW0104+C2402 in Patients With Hypertension and Dyslipidemia
Brief Title: Evaluate the Efficacy and Safety of Co-administration of JW0104+C2402 in Patients With Hypertension and Dyslipidemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JW24301
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JW0104+C2402 (Experimental): JW0104+C2402, 8 weeks, QD (Quaque Die)
  Interventions: Drug: JW0104+C2402
- JW0104+C2403 (Active Comparator): JW0104+C2403, 8 weeks, QD
  Interventions: Drug: JW0104+C2403
- C2402 (Active Comparator): C2402, 8 weeks, QD
  Interventions: Drug: C2402

INTERVENTIONS:
Drug: JW0104+C2402 — For 8 weeks(PO (Per Oral), QD)
  Other Names: NA (Not Applicable)
  Arms: JW0104+C2402
Drug: JW0104+C2403 — For 8 weeks(PO, QD)
  Other Names: NA (Not Applicable)
  Arms: JW0104+C2403
Drug: C2402 — For 8 weeks(PO, QD)
  Other Names: NA (Not Applicable)
  Arms: C2402

SUMMARY:
A Multi-center, Randomized, Double-blind, Parallel, Phase Ⅲ Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of JW0104+C2402 in Patients with Hypertension and Dyslipidemia

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of co-administration of JW0104+C2402 in comparison with co-administration of JW0104+C2403 or C2402 alone in patients with hypertension and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension and dyslipidemia

Exclusion Criteria:

* The subject not meet the specified msBP and LDL-C level

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in msSBP (Systolic Blood Pressure) | week 8
  Check msSBP
Percent change from baseline in LDL-C (Low-Density Lipoprotein Cholesterol) | week 8
  Check LDL-C

SECONDARY OUTCOMES:
change from baseline in msSBP | week 4
  Check msSBP
Change and percent change from baseline in LDL-C | week 4
  Check LDL-C

CONTACTS AND LOCATIONS:
Overall Officials: Minjung Kim, Study Chair — JW Pharmaceutical
Locations (1):
- Gangdong Sacred Heart Hospital, Seoul, South Korea